CLINICAL TRIAL: NCT05979662
Title: Clinical Evaluation of Primary Endoscopic Frontal Sinus Surgery Grade 6 (Draf III) in Patients With Moderate to Severe Eosinophilic Chronic Rhinosinusitis With Polyps
Brief Title: Endoscopic Frontal Sinus Surgery Draf III in Moderate to Severe Eosinophilic Chronic Rhinosinusitis With Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ibrahim Talal Elshamy (Other)
Responsible Party: Sponsor-Investigator, Ibrahim Talal Elshamy, Assistant Lecturer of Otorhinolaryngology, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 34417/1/21
Record Dates: First submitted 2023-07-29; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Endoscopic Frontal Sinus Surgery; Chronic Rhinosinusitis With Nasal Polyps; Draf III; Draf I or IIa

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group one (Experimental): Patients will undergo endoscopic frontal sinus surgery grade 6(Draf III).
  Interventions: Procedure: Endoscopic frontal sinus surgery grade 6(Draf III).
- Group two (Active Comparator): Patients will undergo endoscopic frontal sinus surgery grade 1-3(Draf I or IIa).
  Interventions: Procedure: Endoscopic frontal sinus surgery grade 1-3(Draf I or IIa)

INTERVENTIONS:
Procedure: Endoscopic frontal sinus surgery grade 6(Draf III). — Patients will receive endoscopic frontal sinus surgery grade 6(Draf III).
  Arms: Group one
Procedure: Endoscopic frontal sinus surgery grade 1-3(Draf I or IIa) — Patients will receive endoscopic frontal sinus surgery grade 1-3(Draf I or IIa).
  Arms: Group two

SUMMARY:
The aim of this study is to evaluate the effect of the primary endoscopic frontal sinus surgery on the clinical outcome in patients having moderate to severe eosinophilic chronic rhinosinusitis with polyps with primary outcome measures in form of recurrence of polyp using endoscopic polyp score and Secondary outcome measures include Lund MacKay score, SNOT-22 and need for corticosteroid to control polyp postoperatively.

DETAILED DESCRIPTION:
Chronic rhinosinusitis with nasal polyps (CRSwNP) is a common inflammatory disorder, affecting about 4% of the population worldwide and strongly impacts the quality of life of affected patient.

Eosinophilic chronic rhinosinusitis (ECRS) is a subtype of recalcitrant Chronic rhinosinusitis . Patients with ECRS and generally having a tissue eosinophil >10 cells per high power field (HPF), have worse disease severity and poorer treatment outcomes compared to non-Eosinophilic chronic rhinosinusitis.

ELIGIBILITY:
Inclusion Criteria:

• Patients with moderate or severe eosinophilic chronic rhinosinusitis with polyps who failed appropriate medical treatment in the form of antibiotic, systemic and local corticosteroid for 3 months .

Exclusion Criteria:

* Narrow anteroposterior diameter of frontal sinus ostium(1cm or less)
* Patients showing less or highest degree of radiological complexity of surgery on studying the Computed Tomography.
* Any contraindication for general anesthesia.
* Patients below age of 18 years.
* Incomplete follow up
* previous sinus surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of polyp using endoscopic polyp score | One year postoperatively
  Polyps were evaluated on each side through nasal endoscopy at each visit and graded based on polyp size, resulting in scores of 0 to 4 9. Zero is no polyp, 1 = small polyps in the middle meatus not reaching below the inferior border of the middle turbinate, 2 = polyps reaching below the lower border of the middle turbinate, 3 = large polyps reaching the lower border of the inferior turbinate or polyps medial to the middle turbinate, and 4 = large polyps causing complete obstruction of the inferior nasal cavity. The sum of the left and right nostril scores is the Nasal Polyp Score

SECONDARY OUTCOMES:
Lund MacKay score | One year postoperatively
  The Lund-Mackay staging system scores each sinus (anterior ethmoid, posterior ethmoid, maxillary, frontal, and sphenoid sinuses) according to the following scale: 0 (no opacification), 1 (partial opacification), or 2 (complete opacification).
Sinonasal Outcome Test- 22 | One year postoperatively
  SNOT- 22 was measured based on a 0-5 scale, where 0 defines no problems with the given symptom and 5 defines maximal problems

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Tanta University Hospitals, Tanta, El-Gharbia
  - Tanta University, Tanta, El-Gharbia

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: after the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding autho